CLINICAL TRIAL: NCT06404463
Title: A Phase II Study of Neoadjuvant QL1706 Plus Chemotherapy in Participants With High-Risk ER+/HER2- Early-Stage Breast Cancer (QUEEN-Neo)
Brief Title: QL1706 Plus Chemotherapy as Neoadjuvant Therapy in Early High-Risk ER+/HER2- Breast Cancer
Acronym: QUEEN-Neo
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhimin Shao, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCHBCC-N070
Record Dates: First submitted 2024-05-04; First posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Early Breast Cancer; Neoadjuvant Therapy; HR+HER2- Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Albumin-Bound Paclitaxel; Doxorubicin; Cyclophosphamide; Epirubicin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- QL1706 (Experimental): QL1706 (bispecific antibody (bsAb) targeting PD-1 and CLTA-4)+nab-P-AC/EC
  Interventions: Drug: QL1706 (bispecific antibody targeting PD-1 and CLTA-4); Drug: Albumin-bound paclitaxel; Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Epirubicin

INTERVENTIONS:
Drug: QL1706 (bispecific antibody targeting PD-1 and CLTA-4) — QL1706 is a novel bispecific combination antibody composed of a recombinant humanized IgG4 monoclonal antibody targeting human PD-1 (programmed cell death protein 1) (PSB103) and a recombinant humanized IgG1 monoclonal antibody targeting human CTLA-4 (cytotoxic T-lymphocyte-associated protein 4) (PSB105). Both antibodies have undergone engineering modifications to introduce mutations facilitating their correct assembly and preventing mispairing, and are expressed in the same cell line at a predetermined ratio (approximately 2:1).
Drug: Albumin-bound paclitaxel — Albumin-bound paclitaxel improves the solubility and delivery of paclitaxel to tumor cells by binding to human albumin, facilitating its transportation through the bloodstream and enhancing its uptake into tumor tissue. It works by binding to and stabilizing microtubules within cancer cells, thereby disrupting the normal process of cell division and leading to cell cycle arrest and apoptosis, ultimately resulting in the death of cancer cells.
Drug: Doxorubicin — Doxorubicin, a widely used chemotherapy drug, belongs to the anthracycline class and is effective against various cancers, including breast cancer, leukemia, and sarcomas. It works by intercalating with DNA and inhibiting topoisomerase II, leading to DNA damage and disruption of DNA replication and transcription processes within cancer cells. Despite its efficacy, doxorubicin may cause side effects such as cardiotoxicity and bone marrow suppression, limiting its long-term use in some patients.
Drug: Cyclophosphamide — Cyclophosphamide is a chemotherapy medication commonly used to treat various types of cancers, including lymphoma, leukemia, and breast cancer. It belongs to the class of alkylating agents and works by crosslinking DNA strands, which prevents cell division and leads to cell death. While effective in treating cancer, cyclophosphamide can also cause side effects such as nausea, vomiting, and suppression of the immune system.
Drug: Epirubicin — Epirubicin, a chemotherapy medication, is part of the anthracycline class and is used in the treatment of various cancers, including breast cancer, ovarian cancer, and soft tissue sarcoma. It functions by interfering with DNA replication and RNA synthesis within cancer cells, ultimately leading to cell death. Despite its efficacy, epirubicin can cause side effects such as nausea, hair loss, and bone marrow suppression.

SUMMARY:
This study will look at the efficacy and safety of QL1706 plus albumin-bound paclitaxel followed by AC/EC in a neoadjuvant setting, in high-risk, ER+/HER2- early breast cancer.

DETAILED DESCRIPTION:
This study is a single-arm, single-center, phase II clinical trial aimed at observing and evaluating the effectiveness and safety of QL1706 combined with albumin-bound paclitaxel, sequential AC (doxorubicin/cyclophosphamide) neoadjuvant therapy for early high-risk ER+/HER2- breast cancer.

A total of 76 subjects are planned to be enrolled. After enrollment, subjects will receive QL1706 combined with albumin-bound paclitaxel for 4 cycles followed by sequential AC/EC treatment for 4 cycles. Each treatment cycle will span 3 weeks until the occurrence of a specified treatment termination event, after which subjects will continue to undergo postoperative efficacy and safety assessments.

Safety assessments will be conducted before each QL1706 treatment cycle. Imaging evaluations will be performed every 2 cycles until completion of 8 cycles of treatment to assess efficacy. Additional imaging assessments may be performed as clinically indicated during the study. Tumor imaging assessments will continue until confirmed disease progression according to RECIST v1.1 criteria, initiation of new anti-tumor therapy, withdrawal of consent, or death, whichever occurs first.

Following treatment completion, a treatment completion visit will be conducted. Subjects who discontinue treatment due to reasons other than RECIST v1.1-defined disease progression will undergo regular tumor imaging assessment follow-ups to evaluate time to disease progression. Subjects will also undergo survival follow-up visits every 6 months (every 3 months in the first year and every 6 months thereafter) after treatment completion to collect and record survival status and subsequent anti-tumor treatment information.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily join this study and sign the informed consent form;
2. Female patients aged ≥18 years and ≤70 years old who are newly diagnosed with breast cancer. According to the definition of the latest ASCO/CAP guidelines, histopathologically confirmed ER+/HER2- breast cancer, histological grade II, Ki-67 ≥ 20% and TNM stage T1c-T2, cN1-cN2 or T3- T4, cN0-cN2;
3. According to RECIST 1.1, there is at least one measurable lesion;
4. ECOG score: 0~1;
5. Tumor tissue specimens that can be used for biomarker detection;
6. The function of vital organs meets the following requirements (no blood components or cell growth factor drugs are allowed within 14 days before the first medication):

(1) Absolute neutrophil count ≥1.5×109/L; (2) Platelets ≥100×109/L; (3) Hemoglobin ≥90 g/L; (4) Serum albumin ≥30 g/L; (5) Thyroid-stimulating hormone (TSH) ≤1×ULN (if abnormal, the FT3 and FT4 levels should be examined at the same time. If the FT3 and FT4 levels are normal, you can be included in the group); (6) Serum total bilirubin ≤1.5×ULN; (7) ALT and AST ≤2.5×ULN, if liver metastasis is present, ALT and AST ≤5ULN; (8) AKP≤2.5×ULN; Serum creatinine ≤1.5×ULN; (9) International normalized ratio (INR) ≤1.5 (not receiving anticoagulant therapy).

Exclusion Criteria:

1. The presence of any active autoimmune disease or a history of autoimmune disease (such as the following, but not limited to autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hypophysitis, vasculitis, nephritis, hyperthyroidism; Those who suffer from vitiligo or whose asthma has been completely relieved in childhood and do not need any intervention in adulthood can be included; asthma that requires medical intervention with bronchodilators cannot be included);
2. Are currently using immunosuppressants or systemic hormone therapy to achieve immunosuppression (dose >10 mg/day prednisone or other effective hormones), and are still using it within 2 weeks before enrollment;
3. Severe allergic reactions to other monoclonal antibodies;
4. Known history or evidence of interstitial lung disease or active non-infectious pneumonia;
5. Those with known central nervous system metastasis;
6. Suffered from other malignant tumors in the past 5 years or at the same time (except cured basal cell carcinoma of the skin and cervical cancer in situ);
7. Suffering from high blood pressure that cannot be well controlled by antihypertensive drug treatment (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg); the above parameters are allowed to be achieved through the use of antihypertensive treatment; there has been a hypertensive crisis or high blood pressure in the past Hypertensive encephalopathy;
8. Have cardiac clinical symptoms or diseases that cannot be well controlled, such as (1) NYHA grade 2 or above heart failure (2) Unstable angina (3) Myocardial infarction within 1 year (4) Clinically significant supraventricular infarction or ventricular arrhythmia requiring treatment or intervention (5) QTc>450ms (male); QTc>470ms (female);
9. Those who are receiving thrombolysis or anticoagulation therapy are allowed to use low-dose aspirin and low-molecular-weight heparin prophylactically;
10. Have clinically significant bleeding symptoms or a clear bleeding tendency within 3 months before enrollment; if fecal occult blood is positive during the baseline period, it can be re-examined. If it is still positive after the reexamination, a gastroscopy is required;
11. The tumor invades important blood vessels, or the researcher determines based on imaging that there is a high possibility that the cancer will invade important blood vessels in the future study period, which may lead to fatal bleeding;
12. Patients with pleural effusion, ascites or pericardial effusion that require drainage can be enrolled if the researcher assesses that the symptoms are stable after drainage;
13. Arterial/venous thrombosis events that occurred within 6 months before enrollment, such as cerebrovascular accidents (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism;
14. Known hereditary or acquired bleeding and thrombotic tendencies (such as hemophilia patients, coagulation disorders, etc.);
15. Major vascular disease (for example, aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis) within 6 months before the start of study treatment;
16. Urine routine shows urine protein ≥ ++ and confirmed 24-hour urine protein amount >1.0 g;
17. Suffering from active infection, unexplained fever ≥38.5℃ within 7 days before taking the drug, or baseline white blood cell count >15×109/L;
18. Those with congenital or acquired immune deficiency (such as HIV infection); those who are hepatitis B surface antigen (HBsAg) positive and hepatitis B virus deoxyribonucleic acid (HBV DNA) ≥ 2000 IU/ml, or hepatitis C virus antibody positive;
19. Have received live vaccines less than 4 weeks before study medication or may be vaccinated during the study period;
20. In the judgment of the researcher, the patient has other factors that may affect the study results or cause the study to be terminated midway, such as alcoholism, drug abuse, other serious diseases (including mental illness) that require combined treatment, and serious laboratory tests. Abnormalities, accompanied by family or social factors, may affect the patient's safety.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2024-05-06 (Estimated); Primary Completion 2025-11-06 (Estimated); Study Completion 2030-11-06 (Estimated)

PRIMARY OUTCOMES:
Total Pathological complete response (tpCR) rate using the definition of ypT0/Tis ypN0 | Up to approximately 36 weeks after study start
  No invasive residual in breast or nodes; noninvasive breast residuals allowed ) at the time of definitive surgery

SECONDARY OUTCOMES:
pCR rate using an alternative definition, ypT0/Tis | Up to approximately 36 weeks after study start
  PCR rate (ypT0/Tis) is defined as the percentage of participants without invasive cancer in the breast irrespective of ductal carcinoma in situ or nodal involvement following completion of neoadjuvant systemic therapy by current AJCC staging criteria assessed by the local pathologist at the time of definitive surgery.
pCR rate in PD-L1+ population | Up to approximately 36 weeks after study start
  pCR rate (ypT0/is ypN0) is defined as the percentage of participants without residual invasive on hematoxylin and eosin evaluation of the complete resected breast specimen and all sampled regional lymph nodes following completion of neoadjuvant systemic therapy by current AJCC staging criteria assessed by the local pathologist at the time of definitive surgery in participants with tumors expressing Programmed Death-Ligand 1 (PD-L1).
rate of RCB scored 0-1 | Up to approximately 36 weeks after study start
  Residual cancer burden scored at 0-1 on hematoxylin and eosin evaluation of the complete resected breast specimen and all sampled regional lymph nodes following completion of neoadjuvant systemic therapy assessed by the local pathologist at the time of definitive surgery.
Objective Response Rate (ORR) Objective Response Rate (ORR) Objective Response Rate (ORR) Objective Response Rate (ORR)Objective Response Rate (ORR) | Up to approximately 36 weeks after study start
  ORR is defined as the proportion of participants who have a complete response (CR) or partial response (PR) based on BICR and investigator assessment using RECIST 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Zhimin Shao, MD,PhD, Principal Investigator — Breast cancer institute of Fudan University Cancer Hospital

IPD SHARING:
Plan to Share IPD: No